CLINICAL TRIAL: NCT03314610
Title: Effect of Need to Void on Parkinsonian Gait
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Head of Neuro-Urology Department, Tenon Hospital, Pierre and Marie Curie University
Other Study IDs: P. GREEN 001
Record Dates: First submitted 2017-10-15; First posted 2017-10-19 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Lower Urinary Tract Symptoms; Parkinsonism; Gait Disorders, Neurologic
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Parkinsonian Disorders; Gait Disorders, Neurologic | interventions — Walking Speed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patient with parkinsonian syndromes and lower urinary tract symptoms, age > 18, able to walk without human help on 50 meters, able to hold urine at least 3 minutes. A first record of gait speed will be at strong desire to void. A second record will be after voiding or catheterization Gait records consist on : 3x 10 meter walk test, 1x double task 10 meter walk test, 1x Timed up and Go test and 1x GMT
  Interventions: Other: Gait speed

INTERVENTIONS:
Other: Gait speed — No intervention, only propose water and wait for need to void

SUMMARY:
This study evaluates the effect of the need to void on parkinsonian gait

DETAILED DESCRIPTION:
Parkinsonian syndromes are common causes of gait disorders, associated with hypometria, bradykinesia or rigidity. If motor disorders are the most visible part, lower urinary tract dysfunction is one of the most prevalent dysautonomic disorder (27-80%), especially over active bladder syndrome (OAB). If it seems evident that gait and urinary disorders are linked, because of similar anatomic pathways and control processes, no studies have investigated their association in extrapyramidal patients.

The aim of this study is to assess the effect of the need to void on the walking speed in this particular population.

This prospective study inclues all parkinsonian syndromes who had a follow-up for OAB. They must have a security delay over five minutes, no severe cognitive, motor or psychiatric disorders. We invite them to drink until a need to void (or equivalent). Bladder filling is measured by bladder scan, then they performe gait tests in a specific place, with calm and no passage : Patient can use their habitual walking device. Speed walk asking is comfortable for the two test. Three ten-meter tests, one double-task ten-meter test, one timed-up-and-go test, one timed raise of the floor (GMT). We repeat the same tests after voiding or self-catheterization. Toilets are just next to the hall where they realize the tests. A clinical examination assesses urinary dysfunction (USP, IPSS), motor score (UPDRS-III, Hoehn and Yahr scale, daily equivalent of levodopa), history of falls and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Parkinsonian syndromes
* Follow in neurourology for Lower urinary tract symptoms
* Able to walk 50 meters without human assistance
* able to hold voiding for more than 3 minutes

Exclusion Criteria:

* Actual urinary tract infection
* Montreal cognitive assessment < 20/30
* Acute psychiatric or neurologic disorders who can interfer with walking tests

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in a tertiary center in neuro-urology
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Gait Speed | [Time Frame: 1 Day: at strong desire to void and just after void]
  Gait speed calculated from 10 meter walk test. Time is recorded by a manual chronometer. 3 records are done, mean time is calculated.

SECONDARY OUTCOMES:
Time for Timed up and Go | [Time Frame: 1 Day: at strong desire to void and just after void]
  1 record is done for timed up and go test. Time is recorded by a manual chronometer
Time for GMT | [Time Frame: 1 Day: at strong desire to void and just after void]
  1 record is done for GMT , time is recorded by a manual chronometer
Variation of gait speed | [Time Frame: 1 Day: at strong desire to void and just after void]
  Standard deviation and Coefficient of variation is calculated from the 3 records of 10 meter walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — GREEN GRC-01, Neuro-urology, hôpital Tenon
Locations (1):
- Service de Neuro-urology, hôpital Tenon, Paris, France